CLINICAL TRIAL: NCT02698787
Title: Investigation of the FAST Sound Coding Strategy in Newly Implanted Adult Cochlear Implant Recipients
Brief Title: Fundamental Asynchronous Stimulus Timing Sound Coding Study
Acronym: FAST
Status: Completed | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAM5621
Record Dates: First submitted 2015-12-03; First posted 2016-03-04 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Sensorineural Hearing Loss
Keywords: cochlear implant, sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (2):
- Group 1 (Experimental): All patients will be receiving commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with Contour Advance™ Electrode for this study. Group 1 will be receiving the FAST (experimental) sound coding strategy at initial activation and use it for the first three months.At the three month interval subjects in Group 1 will be switched to the commercially available ACE (control) sound coding strategy.
  Interventions: Device: Experimental sound coding strategy (FAST); Device: Commercially available ACE sound coding strategy
- Group 2 (Experimental): All patients will be receiving commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with Contour Advance™ Electrode for this study. Group 2 will be the commercially available ACE (control) sound coding strategy at initial activation and use it for the first three months.At the three month interval subjects in Group 2 will be switched to the receiving intervention of the FAST (experimental) sound coding strategy. The experimental sound coding strategy will be used from 3-6 months post activation.
  Interventions: Device: Experimental sound coding strategy (FAST); Device: Commercially available ACE sound coding strategy

INTERVENTIONS:
Device: Experimental sound coding strategy (FAST) — Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
Device: Commercially available ACE sound coding strategy — Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy

SUMMARY:
The Fundamental Asynchronous Stimulus Timing (FAST) is a novel cochlear implant sound coding strategy. Potential benefits include improved battery life, in addition to improved localization for bilateral patients.

DETAILED DESCRIPTION:
The Fundamental Asynchronous Stimulus Timing (FAST) strategy offers excellent potential as a low power alternative coding strategy to the current default strategy in Nucleus® cochlear implants, Advanced Combination Encoder (ACE). Additionally, FAST offers potential bilateral benefits - localization and listening in spatially separated noise - because it has been shown in acute, controlled studies to provide more access to interaural timing difference (ITD) cues (Smith, 2010).Previous research with experienced cochlear-implant recipients has shown issues with conversion from ACE to FAST. The FAST strategy typically sounds very different in quality, and acclimatization can be lengthy. This extended adaptation time makes it difficult to show conclusively that FAST is non-inferior to ACE for speech understanding. A potential barrier to evaluating performance with FAST in current cochlear-implant recipients is the extensive amount of prior experience that many recipients have using ACE. Hence, there is a distinct need to evaluate FAST in newly implanted recipients.

ELIGIBILITY:
Inclusion Criteria

* Medical and audiological candidate for a unilateral CI24RE, CI512 or CI532 series implant
* Post-linguistically deafened
* Native speaker of American English
* Eighteen years of age or older

Exclusion Criteria

* Previous or existing cochlear-implant recipient
* Pre-linguistically deafened (onset of hearing loss at less than two years of age)
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Diagnosis of retro-cochlear pathology
* Diagnosis of auditory neuropathy
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and use of the prosthetic device
* Unwillingness or inability to comply with all investigational requirements
* Additional cognitive handicaps that would delay rate of improvement with the cochlear implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Health, Aurora, Colorado, United States

REFERENCES:
- [Background] Daneman , M., & Carpenter, P.A. (1980). Individual differences in working memory and reading. Journal of Verbal Learning andVerbal Behavior, 19, 450-466.
- [Background] Noble W, Jensen NS, Naylor G, Bhullar N, Akeroyd MA. A short form of the Speech, Spatial and Qualities of Hearing scale suitable for clinical use: the SSQ12. Int J Audiol. 2013 Jun;52(6):409-12. doi: 10.3109/14992027.2013.781278. PMID 23651462
- [Background] Bench J, Kowal A, Bamford J. The BKB (Bamford-Kowal-Bench) sentence lists for partially-hearing children. Br J Audiol. 1979 Aug;13(3):108-12. doi: 10.3109/03005367909078884. PMID 486816
- [Background] PETERSON GE, LEHISTE I. Revised CNC lists for auditory tests. J Speech Hear Disord. 1962 Feb;27:62-70. doi: 10.1044/jshd.2701.62. No abstract available. PMID 14485785
- [Background] Smith, Z. M. (2010). Improved sensitivity to interaural time differences with the FAST coding strategy. Presented at the 11th International Conference on Cochlear Implants and Other Implantable Auditory Technologies, Stockholm, Sweden.

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: FAST First, Then ACE Sound Coding Strategy: All patients will be receiving commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with Contour Advance™ Electrode for this study. Group 1 will be receiving the FAST (experimental) sound coding strategy at initial activation and use it for the first three months.At the three month interval subjects in Group 1 will be switched to the commercially available ACE (control) sound coding strategy.
  Experimental sound coding strategy (FAST): Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
  Commercially available ACE sound coding strategy: Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
- Group 2: ACE First, Then FAST Sound Processng Strategy: All patients will be receiving commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with Contour Advance™ Electrode for this study. Group 2 will be the commercially available ACE (control) sound coding strategy at initial activation and use it for the first three months.At the three month interval subjects in Group 2 will be switched to the receiving intervention of the FAST (experimental) sound coding strategy. The experimental sound coding strategy will be used from 3-6 months post activation.
  Experimental sound coding strategy (FAST): Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
  Commercially available ACE sound coding strategy: Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
Period: First Intervention (3 Months)
Arm/Group | Group 1: FAST First, Then ACE Sound Coding Strategy | Group 2: ACE First, Then FAST Sound Processng Strategy
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention (3 Months)
Arm/Group | Group 1: FAST First, Then ACE Sound Coding Strategy | Group 2: ACE First, Then FAST Sound Processng Strategy
Started | 6 | 5
Completed | 6 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: FAST First, Then ACE Sound Processing Strategy: All patients will be receiving commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with Contour Advance™ Electrode for this study. Group 1 will be receiving the FAST (experimental) sound coding strategy at initial activation and use it for the first three months.At the three month interval subjects in Group 1 will be switched to the commercially available ACE (control) sound coding strategy.
  Experimental sound coding strategy (FAST): Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
  Commercially available ACE sound coding strategy: Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
- Group 2: ACE First, Then FAST Sound Processing Strategy: All patients will be receiving commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with Contour Advance™ Electrode for this study. Group 2 will be the commercially available ACE (control) sound coding strategy at initial activation and use it for the first three months.At the three month interval subjects in Group 2 will be switched to the receiving intervention of the FAST (experimental) sound coding strategy. The experimental sound coding strategy will be used from 3-6 months post activation.
  Experimental sound coding strategy (FAST): Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
  Commercially available ACE sound coding strategy: Commercially available Cochlear™ Nucleus® CI24RE with Contour Advance™ Electrode or Cochlear™ Nucleus® CI512 cochlear implant with FAST sound coding strategy using crossover design in newly implanted subjects. Both groups will receive the experimental and control strategy
- Total: Total of all reporting groups
Arm/Group | Group 1: FAST First, Then ACE Sound Processing Strategy | Group 2: ACE First, Then FAST Sound Processing Strategy | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Full Range); unit: years] | 66.4 [33.3 to 78.1] | 54.36 [22.7 to 79.4] | 60.9 [22.7 to 79.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Open Set Monosyllabic Word Recognition Score
Description: Open Set Monosyllabic Word Recognition is a test of 50 words each consisting of 3 individual speech sounds. The subject repeats the word s/he hears to the audiologist. The score is based on the percentage of words correct.
  The primary outcome measure to is determine if the investigational sound coding strategy (FAST) is non-inferior to commercially approved sound coding strategies (ACE) for word recognition in quiet with percentage of words correct.
Time Frame: Visit 1 (baseline), Visit 5 (3 months), Visit 8 (6 months)
Population: Group 1 were analysed at Visit 5 for FAST sound coding strategy and at Visit 8 for ACE sound coding strategy. Group 2 were analysed at Visit 5 for ACE sound coding strategy and at Visit 8 for FAST sound coding strategy.
Measure: Mean (Full Range); unit: percentage of words correct
Arm/Group | Group 1: FAST First, Then ACE Sound Processing Strategy | Group 2: ACE First, Then FAST Sound Processing Strategy
Number analyzed (Participants) | 6 | 5
percentage of words correct
  Visit 1 (Candidacy) - Implated Ear | 5 [0 to 17] | 11.8 [0 to 27]
  Visit 1 (Candidacy) - Contralateral Ear | 20.2 [1 to 55] | 21.4 [2 to 38]
  Visit 5 (3 Months) - FAST: number analyzed (Participants) | 6 | 0
  Visit 5 (3 Months) - FAST | 45 [9 to 69] |
  Visit 5 (3 Month) - ACE: number analyzed (Participants) | 0 | 5
  Visit 5 (3 Month) - ACE |  | 59.4 [39 to 85]
  Visit 8 (6 Month) - ACE: number analyzed (Participants) | 6 | 0
  Visit 8 (6 Month) - ACE | 49.5 [15 to 79] |
  Visit 8 (6 Month) - FAST: number analyzed (Participants) | 0 | 4
  Visit 8 (6 Month) - FAST |  | 54 [27 to 76]

2. Primary Outcome: Change in Signal-to-Noise Ratio (SRT)
Description: The primary outcome measure to is determine if the investigational sound coding strategy (FAST) is non-inferior to commercially approved sound coding strategies (ACE) for BKB sentences in noise with mean signal-to-noise ratio (SRT) where participants could understand 50% of sentences in noise using ACE and FAST. Lower SRT values indicate better performance.
  SRT measures are obtained using two types of background noise. One is "Speech-Shaped Noise" which is white noise or tones made to mimic speech. The other is "Four-Talker Noise" which is multiple talkers made to mimic background conversation.
Time Frame: Visit 5 (3 Months) and Visit 8 (6 months)
Population: as for outcome 1
Measure: Mean (Full Range); unit: signal-to-noise ratio
Arm/Group | Group 1: FAST First, Then ACE Sound Processing Strategy | Group 2: ACE First, Then FAST Sound Processing Strategy
Number analyzed (Participants) | 6 | 5
signal-to-noise ratio
  Visit 5 - FAST (Speech-Shaped Noise): number analyzed (Participants) | 6 | 0
  Visit 5 - FAST (Speech-Shaped Noise) | 16.3 [9.1 to 32.6] |
  Visit 5 - FAST (Four-Talker Noise): number analyzed (Participants) | 6 | 0
  Visit 5 - FAST (Four-Talker Noise) | 16.3 [7.8 to 30.5] |
  Visit 5 - ACE(Speech-Shaped Noise): number analyzed (Participants) | 0 | 5
  Visit 5 - ACE(Speech-Shaped Noise) |  | 11.2 [4.9 to 21.6]
  Visit 5 - ACE (Four-Talker Noise): number analyzed (Participants) | 0 | 5
  Visit 5 - ACE (Four-Talker Noise) |  | 10.1 [4.1 to 23.0]
  Visit 8 - FAST (Speech-Shaped Noise): number analyzed (Participants) | 0 | 4
  Visit 8 - FAST (Speech-Shaped Noise) |  | 13.1 [5.8 to 28.0]
  Visit 8 - FAST (Four-Talker Noise): number analyzed (Participants) | 0 | 4
  Visit 8 - FAST (Four-Talker Noise) |  | 12.4 [7 to 26]
  Visit 8 - ACE(Speech-Shaped Noise): number analyzed (Participants) | 6 | 0
  Visit 8 - ACE(Speech-Shaped Noise) | 9.9 [6.1 to 14.8] |
  Visit 8 - ACE (Four-Talker Noise): number analyzed (Participants) | 6 | 0
  Visit 8 - ACE (Four-Talker Noise) | 9.1 [6.0 to 15.9] |

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events are categorized by the intervention used at the time of adverse event onset. All subjects received a commercially available cochlear implant and then took a resting period of approximately two weeks prior to starting ACE or FAST sound coding strategies. It is common for all cochlear implant recipients to experience adverse events during or after surgery. Adverse events which occur prior to starting a sound coding strategy are listed under "No Sound Coding Strategy".
Groups:
- No Sound Coding Strategy: Healing period after surgery.
- FAST Sound Coding Strategy: Participants utilising the FAST Sound Coding Strategy. Group 1 utilises in first 3 months, Group 2 utilises in second 3 months.
- ACE Sound Coding Strategy: Participants utilising the ACE Sound Coding Strategy. Group 1 utilises in second 3 months, Group 2 utilises in first 3 months.
Arm/Group | No Sound Coding Strategy | FAST Sound Coding Strategy | ACE Sound Coding Strategy
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 5/11 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Sound Coding Strategy (N=11) | FAST Sound Coding Strategy (N=11) | ACE Sound Coding Strategy (N=11)
Vertigo/dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Sound Coding Strategy (N=11) | FAST Sound Coding Strategy (N=11) | ACE Sound Coding Strategy (N=11)
"Whooziness" (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear canal scaly and slightly swollen (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Profound hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — Sudden hearing threshold shift
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0)
Unsteadiness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Disabled E12 (Product Issues) | 0 (0) | 1 (1) | 0 (0) — Poor sound quality and perception
Cerebrospinal fluid release (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Resolved during surgery
Vertigo and dizziness (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent non-auditory stimulation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Non-auditory stimulator (Product Issues) | 0 (0) | 1 (1) | 0 (0) — Disabled electrode
Change in sound quality (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Impedance spiked (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Change in audibility (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Tenderness around device (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Non-auditory sensation/pain (Product Issues) | 0 (0) | 1 (1) | 0 (0) — Disabled electrode
Disabled electrode 14 following pitch ranking (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Intermittent sound (Product Issues) | 0 (0) | 2 (2) | 0 (0)
Disabled E22 (Product Issues) | 0 (0) | 1 (1) | 0 (0) — Sound quality and significantly higher threshold and comfort levels
Redness and Indentation at magnet site (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Significant increase in impedances (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Worsening sinus symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Short circuit electrode(s) (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Electrode tip roll/fold-over (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Swelling and slight soreness/sensitivity around internal device (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Lethargic (General disorders) | 1 (1) | 0 (0) | 0 (0)
Soreness on posterior border of implant (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Low-grade headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT02698787/Prot_SAP_000.pdf